CLINICAL TRIAL: NCT05081427
Title: Non-invasive Biomarkers of Metabolic Liver Disease (NIMBLE); An FNIH Biomarkers Consortium Study: Study 1.2
Brief Title: Non-invasive Biomarkers of Metabolic Liver Disease (NIMBLE) Study 1.2
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Foundation for the National Institutes of Health (Other)
Responsible Party: Principal Investigator, Sudhakar K. Venkatesh, M.D., Principal Investigator, Mayo Clinic
Other Study IDs: 20-012529
Record Dates: First submitted 2021-10-06; First posted 2021-10-18 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Nonalcoholic Fatty Liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a prospective, observational, single-center, short-term cross-sectional study to assess the repeatability and reproducibility of a set of specified MRI quantitative biomarkers.

DETAILED DESCRIPTION:
NIMBLE is a comprehensive, five-year collaborative effort to standardize, compare, validate, and advance the regulatory qualification of imaging and circulating biomarkers to diagnose and stage nonalcoholic steatohepatitis (NASH), and to predict and assess response to therapeutic intervention (https://fnih.org/what-we-do/biomarkers-consortium/programs/nimble).

The purpose of this study is to assess the repeatability and reproducibility of a set of specified MRI quantitative biomarkers. The imaging biomarkers will cover an array of methods that could be applicable to non-alcoholic fatty liver disease (NAFLD), including liver fat, liver stiffness, corrected T1 relaxation time and body composition assessments. The data collected will be used to inform a decision of which of these biomarkers has sufficient precision to be advanced to NIMBLE Stage 2.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age ≥ 18 years).
* Known or suspected NAFLD based on:
* Prior biopsy ≤ 36 months consistent with NAFLD; OR
* Clinical and laboratory data ≤ 3 months before enrollment consistent with NAFLD: abnormal ALT (>30 U/L for men, > 19 U/L for women) without other common causes such as HCV, HBV AND meets criteria or ATP III criteria (2005 revision) for metabolic syndrome with any 3 of the 5:

  i. Waist circumference (WC) > 102 cm (M) or > 88 cm (F) ii. Fasting glucose ≥ 100 mg/dL or Rx iii. TG ≥ 150 mg/dL or Rx iv. Elevated blood pressure (SBP ≥ 130 mmHg or DBP ≥ 85 mmHg) v. Reduced HDL-C < 40 mg/dL (M) or < 50 gm/dL (W)
* Able and willing to participate, including maintaining steady-state: diet, physical activity, alcohol use, medications.
* Classifiable into one of the following enrollment categories by FIB-4 (ALT, AST, platelets, date of birth) collected at screening visit if not available already within 3 months prior:
* Low likelihood of advanced fibrosis: FIB-4 ≤ 1.3 (about one-third of enrolled subjects, minimum 20%, maximum 45%);
* Intermediate likelihood of advanced fibrosis: 1.3 < FIB-4 < 2.67 (about one-third of enrolled subjects, minimum 20%, maximum 45%);
* High likelihood of advanced fibrosis: FIB-4 ≥ 2.67: (about one-third of enrolled subjects, minimum 20%, maximum 45%).

Exclusion Criteria:

1. Liver disease other than NAFLD
2. Excess alcohol consumption (≥ 2 units/day for women and ≥ 3 units/day for men)
3. Current diagnosis of drug induced liver injury
4. Receiving drug or placebo in treatment trial now or within 30 days
5. Weight loss or gain of ≥ 5 kg in prior 3 months
6. Other factors that in the judgment of the PI might preclude study completion
7. Women who state they are pregnant. Women who state they are pregnant will be excluded in an abundance of caution, since pregnancy might increase intra-abdominal pressure which in turn might affect the assessment of the different-day reproducibility coefficient of MRI and VCTE measurements.
8. Patients with active implants such as pacemakers or defibrillators or any other contraindication to MRI or VCTE scanning.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective cross-sectional study will enroll subjects 18 years or older with suspected or confirmed diagnosis of NAFLD. Based on protocol-specified FIB-4 values, about one-third are expected to have low, one-third to have intermediate, and one-third to have high likelihood of advanced fibrosis.
  The study will use an interim analysis, adaptive MRI protocol, and adaptive sample size. It is anticipated that up to a total of 48 subjects will be enrolled and complete imaging protocols.
  General health status: Patients with suspected or confirmed diagnosis of NAFLD and no contraindications for an MRI exam.
  Geographic location: Rochester, Minnesota
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Reproducibility of liver stiffness | Within 7 days
  Repeatability liver stiffness in kilopascals (kPa)
Reproducibility of liver fat content | Within 7 days
  Repeatability of liver proton density fat fraction (PDFF) in %
Reproducibility of visceral adipose tissue volume | Within 7 days
  Repeatability of visceral adipose tissue volume measured in mL

CONTACTS AND LOCATIONS:
Overall Officials: Sudhakar Venkatesh, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Fowler KJ, Venkatesh SK, Obuchowski N, Middleton MS, Chen J, Pepin K, Magnuson J, Brown KJ, Batakis D, Henderson WC, Shankar SS, Kamphaus TN, Pasek A, Calle RA, Sanyal AJ, Loomba R, Ehman R, Samir AE, Sirlin CB, Sherlock SP. Repeatability of MRI Biomarkers in Nonalcoholic Fatty Liver Disease: The NIMBLE Consortium. Radiology. 2023 Oct;309(1):e231092. doi: 10.1148/radiol.231092. PMID 37815451
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials